CLINICAL TRIAL: NCT05420896
Title: Electromyographic Evaluation of the Efficacy of Manual Therapy in Temporomandibular Joint
Brief Title: Electromyographic Evaluation of the Efficacy of Manual Therapy in Temporomandibular Joint Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Kumru Ateş, PhD-C, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BahçesehırÜniversitesi
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Temporomandibular Joint Dysfunction
Keywords: temporomandibular joint dysfunction; manual therapy; EMG; maximal mouth opening
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy (Active Comparator): Upper cervical spine mobilization Posterior-anterior mobilization of the fifth cervical vertebra Suboccipital inhibition Suboccipital mobilization Trigger point application to my masseter, temporal and sternocleidomastoid muscles Intraoral and extraoral myofascial release Intraoral sphenopalatine ganglion technique TMJ mobilization Massage for chewing muscles The 45-minute treatment program, which includes applications including the techniques above, will be applied to the patients randomly assigned to the study group once a week for a total of 4 weeks.The changes in muscle activity of the masseter and anterior temporalis bilaterally will be recorded with EMG.
  Interventions: Other: Manual Therapy
- Control group (No Intervention): Patients assigned to the control group randomly will be re-evaluated 4 weeks after their initial evaluation. No intervention will be applied during this period. After 4 weeks, when the patients are re-evaluated, they will be directed to the appropriate treatment.

INTERVENTIONS:
Other: Manual Therapy — Upper cervical spine mobilization Posterior-anterior mobilization of the fifth cervical vertebra Suboccipital inhibition Suboccipital mobilization Trigger point application to my masseter, temporal and sternocleidomastoid muscles Intraoral and extraoral myofascial release Intraoral sphenopalatine ganglion technique TMJ mobilization Massage for chewing muscles The 45-minute treatment program, which includes applications including the techniques above, will be applied to the patients randomly assigned to the study group once a week for a total of 4 weeks.The changes in muscle activity of the masseter and anterior temporalis bilaterally will be recorded with EMG.
  Arms: Manual therapy

SUMMARY:
Individuals with temporomandibular joint dysfunction (TMD) may experience changes in muscle activation as a result of symptoms such as pain and limitation of movement. The aim of this study is to examine the efficacy of manual therapy electromyographically in patients with TMD.

DETAILED DESCRIPTION:
TMD is a common condition in the community. It may occur due to factors such as trauma, stress, occlusal disorders. Symptoms include pain, limitation in mouth opening, joint voice, postural and psychosocial disorders. TMD/RDC diagnostic criteria are used in the classification of TMD, and accordingly, it is stated that it may originate from the joint, disc and chewing muscles. In the treatment, conservative treatments such as patient education, manual therapy and exercises are applied first.

Manual therapy is an effective physiotherapy method on pain and muscle dysfunctions in musculoskeletal problems. In our study, electromyographic changes of masticatory muscles will be examined by applying manual treatment to the masticatory muscles and cervical region in myofascial TMD patients according to TMD/RC.

ELIGIBILITY:
Inclusion Criteria:

* No cognitive impairment
* Diagnosed with temporomandibular joint(TMJ) dysfunction of myofascial origin,
* Volunteers aged 18-65

Exclusion Criteria:

* Malignancy and fracture of the cervical region and/or TMJ
* Active infection
* Patients actively receiving cervical and/or TMJ-related therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from initial assessment to 4 weeks after initial assessment.
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.

SECONDARY OUTCOMES:
Electromyography (EMG) | Change from initial assessment to 4 weeks after initial assessment.
  Electromyography (EMG) is the most objective and reliable method available for imaging muscle function and efficiency, which is done by identifying their electrical potentials. In global surface electromyography (sEMG), surface electrodes are located on the surface of the skin, and it detects superimposed motor unit action potentials from many muscle fibers
Pain Pressure Threshold (PPT) | Change from initial assessment to 4 weeks after initial assessment.
  Pain pressure threshold (PPT) is used to measure deep muscular tissue sensitivity. The test determines the amount of pressure over a given area in which a steadily increasing nonpainful pressure stimulus turns into a painful pressure sensation. A varying pressure is applied from 0.5 to 1 kg/sec in a perpendicular direction relative to the muscle.
Maximum Mouth Opening (MMO) | Change from initial assessment to 4 weeks after initial assessment.
  Maximal opening of mouth is described as the greatest distance between incisal edge of maxillary central incisor to the incisal edge of mandibular central incisor, when the mouth is opened as wide as possible painlessly or as the inter incisal distance plus the overbite. Clinical measurement of normal range of Maximum Mouth Opening (MMO) is an important diagnostic criterion for evaluation of stomatognathic system, especially for those with temporomandibular dysfunctions.
TAMPA | Change from initial assessment to 4 weeks after initial assessment.
  The original Tampa Scale of Kinesiophobiais (TSK) was first developed in 1991 by R. Miller, S. Kopri, and D. Todd. TSK is 12 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance.
  The questionnaire using 4 points to assess that are based on; the model of fear-avoidance, fear of work-related activities, fear of movement, and fear of re-injury.
Functional Limitation Scale of the Jaw-8 | Change from initial assessment to 4 weeks after initial assessment.
  It is a scale used to evaluate the functionality of the individual's jaw joint in the last month. It consists of 8 items, where the number '0' indicates 'no restriction' and the number '10' indicates 'serious restriction'. By taking the average of the answers given, the functionality restriction is calculated.
Hospital Anxiety Depression Scale (HADS) | Change from initial assessment to 4 weeks after initial assessment.
  The Hospital Anxiety Depression Scale (HADS) includes two subscales, seven of which measure anxiety (odd numbers) and seven (even numbers) depression, which are used to determine the depression and anxiety levels of individuals, and a total of 14 questions. Each question is scored between 0-3 points. While the minimum score that can be obtained from the depression and anxiety subscales is 0, the maximum score is 21. According to the scores obtained from the subscales, the depression and anxiety status of the individuals are evaluated as normal/no symptoms (0-7 points), borderline abnormal/suspicious (8-10 points), and abnormal/definite (11-21 points).

CONTACTS AND LOCATIONS:
Overall Officials: Kumru Ateş, PhC, Principal Investigator — Bahçeşehir University
Locations (1):
- Bahçeşehir University, Istanbul, Europe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No